CLINICAL TRIAL: NCT04062370
Title: Different Regimens of Ranibizumab Treatment for Macular Edema Secondary to Retinal Vein Occlusion: a Randomized and Controlled Clinical Study.
Brief Title: Ranibizumab Treatment for Macular Edema Secondary to Retinal Vein Occlusion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Chen-jin, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019KYPJ092
Record Dates: First submitted 2019-07-29; First posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Retinal Vein Occlusion; Treatment; Photocoagulation Burn to Retina; Ranibizumab
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Ranibizumab

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, controlled, parallel, open-label, exploratory clinical trial. Including 100 patients, 50 : 50 in each arm. Different frequency of Ranibizumab is applied in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1+PRN (Experimental): Intravitreal injection of Ranibizumab 0.5 mg (IVR): initial injection for 1 time ( month 1), and then IVR is required if central macular thickness (CMT) greater than 300 μm during the follow-up observation (Pro re nata, PRN, means if necessary).
  After 6 months follow-up, patients in this arm will be randomly divided to receive IVR PRN only or laser photocoagulation combined with IVR PRN.
  IVR PRN only: patient will receive IVR PRN if CMT greater than 300 μm during the follow-up observation (PRN) after month 6.
  Laser photocoagulation with IVR PRN: patient will receive laser photocoagulation for non-perfusion area according to FFA results after month 6, and then received IVR PRN if CMT greater than 300 μm.
  Interventions: Drug: Ranibizumab; Device: laser photocoagulation
- 3+PRN (Active Comparator): Intravitreal injection of Ranibizumab 0.5 mg (IVR): initial injection for 3 consecutive times ( months 1, 2 and 3 ),and then IVR is required if CMT greater than 300 μm during the follow-up observation (PRN).
  After 6 months follow-up, patients in this arm will be randomly divided to receive IVR PRN only or laser photocoagulation combined with IVR PRN.
  IVR PRN only: patient will receive IVR PRN if CMT greater than 300 μm during the follow-up observation (PRN) after month 6.
  Laser photocoagulation with IVR PRN: patient will receive laser photocoagulation for non-perfusion area according to FFA results after month 6, and then received IVR PRN if CMT greater than 300 μm.
  Interventions: Drug: Ranibizumab; Device: laser photocoagulation

INTERVENTIONS:
Drug: Ranibizumab — Patients will receive intravitreal injection of Ranibizumab 0.5 mg (1+PRN or 3+PRN) according to the study until month 6. Then, patients will received Ranibizumab PRN only or laser photocoagulation with Ranibizumab PRN after month 6.
  Other Names: Lucentis
Device: laser photocoagulation — After month 6, patients will received Ranibizumab PRN only or laser photocoagulation with Ranibizumab PRN according the re-randomization at month 6.

SUMMARY:
Retinal vein occlusion (RVO) may lead to series of complications including retinal ischemia, macular edema (ME) and induce vision impairment. Intravitreal injection of Ranibizumab (0.5mg) has been proved to be a safe and effective method for the treatment of RVO-ME. In this study, different treatment regimens of Ranibizumab is applied and the effects is observed at 1-6 months to explore the best regimen for RVO. After 6 months, anti-VEGF therapy and/or laser photocoagulation is used to explore whether laser photocoagulation can maintain the therapeutic effect of Ranibizumab or reduce the injection number.

DETAILED DESCRIPTION:
Retinal vein occlusion (RVO) may lead to series of complications including retinal ischemia, macular edema (ME) and so on. Retinal vein occlusion (RVO) can be classified as branch retinal vein occlusion (BRVO) and central retinal vein occlusion (CRVO). Retinal vein occlusion with macular edema (RVO-ME) is the main cause of RVO induced vision impairment. Intravitreal injection of Ranibizumab (0.5mg) has been proved to be a safe and effective method for the treatment of RVO-ME. Although multiple injections of anti-vascular endothelial growth factor (anti-VEGF) drugs are beneficial to the therapeutic results of RVO-ME, they may also increase the risk of systemic or ocular complications and at the same time increase the economic burden of patients to a certain extent. Different studies have shown that anti-VEGF therapy with low frequency injection (2-5 doses) is also effective for RVO-related ME. However, there are still different views on which option is better. Meanwhile, the effect of laser photocoagulation in the non-perfusion area of the retina, and whether the number of subsequent anti-VEGF injections can be reduced accordingly, is still uncertain. Therefore, in this study, different treatment regimens will be applied and the effects will be observed at 1-6 months. After 6 months, anti-VEGF therapy and/or laser photocoagulation will be used to explore whether laser photocoagulation can maintain the therapeutic effect or reduce the injection number of Ranibizumab. This study intends to explore the therapeutic effects of different treatment regimens on RVO-ME, and meanwhile to investigate the dynamic changes in retinal morphology, microcirculation and visual function during RVO treatment by means of angiography-optical coherence tomography (angio-OCT), microperimetry, electroretinogram (ERG) examination and other methods.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with RVO-ME diagnosed definitely by FFA and OCT, with CMT > 300μm; BCVA from 20/200 to 20/40 (including 20/200 and 20/40), with a degree of myopia ≤-6 diopter (diopter, D);
2. Patients with a course of RVO ≤ 12 weeks; Patients who have not received laser, intraocular or systemic anti-VEGF treatments or long-acting hormone intraocular, periocular or systemic treatments since the onset of RVO;
3. Patients who are voluntary to sign and date the informed consent form approved by the Ethics Review Committee prior to the conduct of the relevant study steps.

Exclusion Criteria:

1. Patients with a course of disease > 12 weeks;
2. Patients treated with any anti-angiogenic medicines for either eye within 3 months before the baseline; or patients currently in treatment with systemic anti-angiogenic drugs;
3. Patients with their study eyes treated with panretinal photocoagulation (PRP) previously;
4. Patients previously participating in other clinical trials 3 months before the baseline;
5. Patients with severely opacity of refractive media affecting laser treatment and observation;
6. Patients with other ophthalmic diseases affecting visual prognosis, such as corneal disease, glaucoma, severe cataract, uveitis, other fundus diseases, etc.
7. Patients with in any condition where intravitreal injection is unacceptable;
8. Patients identified by the investigator to be medically or mentally unstable: complicated with cardiovascular, cerebrovascular, liver, kidney and hematopoietic system and other serious primary diseases or mental disease; Women who are pregnant or preparing for pregnancy or in lactation, etc.
9. Patients with any history may interfere with the results of the trial or increase the risk of the patient (assessed by the investigator) ;
10. Patients who are in poor compliance and unable to strictly implement the protocol (assessed by the investigator).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
best-corrected visual acuity (BCVA) at month 6 | Month 6 after first treatment
  best-corrected visual acuity (BCVA) at month 6
Central macular thickness (CMT) at month 6 (3) the number of intravitreal injections of Ranibizumab at month 6 | Month 6 after first treatment
  Central macular thickness (CMT) at month 6
the number of intravitreal injections of Ranibizumab at month 6 | Month 6 after first treatment
  the number of intravitreal injections of Ranibizumab at month 6

SECONDARY OUTCOMES:
best-corrected visual acuity (BCVA) at month 12 | Month 12 after first treatment
  best-corrected visual acuity (BCVA) at month 12
the number of intravitreal injections of Ranibizumab at month 12 | Month 12 after first treatment
  the number of intravitreal injections of Ranibizumab at month 12

OTHER OUTCOMES:
best-corrected visual acuity (BCVA) during the follow-up | during the follow-up for up to 12 months.
  best-corrected visual acuity (BCVA) during the follow-up
intraocular pressure during the follow-up | during the follow-up for up to 12 months.
  intraocular pressure during the follow-up
central macular thickness during the follow-up | during the follow-up for up to 12 months.
  central macular thickness during the follow-up
posterior choroidal thickness during the follow-up | during the follow-up for up to 12 months.
  posterior choroidal thickness during the follow-up
The results of angio-optical coherence tomography (angio-OCT) examination during the follow-up | during the follow-up for up to 12 months.
  The results of angio-OCT examination, including area of non-perfusion and neovascularization.
Fundus fluorescein angiography (FFA) examination results during the follow-up | during the follow-up for up to 12 months.
  FFA examination results during the follow-up, including area of non-perfusion and neovascularization.
Microperimetry during the follow-up | during the follow-up for up to 12 months.
  Changes in posterior pole found by microperimetry
Electroretinogram (ERG) during the follow-up | during the follow-up for up to 12 months.
  Amplitudes and implicit times of the a wave and b wave of ERG during the follow-up
adverse events occurring in the follow-up | during the follow-up for up to 12 months.
  Records of adverse events occurring in the follow-up period: including subconjunctival hemorrhage, infection, increased intraocular pressure, retinal tear, retinal detachment, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Chenjin Jin, Ph.D, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Chuangxin Huang, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Campochiaro PA, Hafiz G, Mir TA, Scott AW, Solomon S, Zimmer-Galler I, Sodhi A, Duh E, Ying H, Wenick A, Shah SM, Do DV, Nguyen QD, Kherani S, Sophie R. Scatter Photocoagulation Does Not Reduce Macular Edema or Treatment Burden in Patients with Retinal Vein Occlusion: The RELATE Trial. Ophthalmology. 2015 Jul;122(7):1426-37. doi: 10.1016/j.ophtha.2015.04.006. Epub 2015 May 9. PMID 25972260